CLINICAL TRIAL: NCT01623206
Title: Prospective, Open-labelled, Phase II Study, of the Administration of Desmopressin in Patients With Colorectal Cancer, With or Without Metastasis, With Rectal Bleeding, Before Treatment With Surgery and/or Chemotherapy and/or Radiotherapy.
Brief Title: Desmopressin (DDAVP) in Patients With Colorectal Cancer and Rectal Bleeding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DDAVP-R01-02
Record Dates: First submitted 2012-05-28; First posted 2012-06-19 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Cancer; Rectal Bleeding
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Hemorrhage | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desmopressin (Experimental): Four dose levels and two dosing schedules with 3 patients in each group.
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — Dose groups: Group 1: 0.25 µg/kg/day; Group 2: 0.25 µg/kg/12 hours; Group 3: 0.50 µg/kg/12 hours; Group 4: 1 µg/kg/day; Group 5: 1 µg/kg/12 hours; Group 6: 2 µg/kg/day.
  All groups will receive desmopressin intravenously, in a 15-20 minutes infusion, one or two times a day. The administration will be repeated 24 hours after the first infusion.

SUMMARY:
The objective of this study is to find the maximum tolerated dose and preliminary efficacy of desmopressin as an haemostatic agent, when is administered to patients with colorectal cancer and rectal bleeding, before specific oncologic treatment with surgery and/or chemotherapy and/or radiotherapy.

DETAILED DESCRIPTION:
Colorectal cancer is the third cause of cancer in men and women, according to data recently published in the United Sates, and the third cause of death in the same population. Ninety percent (90%) of patients have symptoms at the time of diagnosis, being rectal bleeding the most frequent one (50% of cases). Bleeding, mainly mild or moderate, has no specific treatment, and during the staging of the disease, can not be controlled.

Desmopressin, a synthetic analogue of vasopressin, is a selective agonist of the receptor V2 of vasopressin, inducing, among others, an haemostatic effect. Interestingly, the expression of this receptor has been described in human gastrointestinal tract, including colon and rectum and in colorectal tumors. Moreover, desmopressin has shown a significant antitumor activity in preclinical murine models of colorectal cancer.

This is a dose finding study, to investigate a new indication of desmopressin as an haemostatic agent in patients with colorectal cancer with mild to moderate rectal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 to < 80 years of age who have signed the informed consent form
* Histological diagnosis of rectal adenocarcinoma localized, locally advanced or metastatic
* Treatment indication with chemotherapy and/or radiotherapy and/or surgery according to disease stage
* Rectal bleeding associated with the primary tumor within 48 hours prior to study entry
* Acceptable organ function to be able to participate in the study, performed within 14 days prior to admission; defined by the following parameters:

  * Electrocardiogram (ECG) without significant clinical abnormalities
  * Haemoglobin greater than or equal to 8 g/dL
  * Total leukocyte count greater than or equal to 4.0 x 10^9/L
  * Absolute neutrophil count greater than or equal to 1.5 x 10^9/L
  * Total platelet count greater to 100.0 x 10^9/L
  * Total bilirubin less than or equal to 1.5 times the upper limit of normality (ULN)
  * Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) less than or equal to 1.5 times upper limit of normality (ULN)
  * Creatinine clearance greater than 50 ml/min
* Performance status (Eastern Cooperative Oncology Group [ECOG]) less than or equal to 2
* Patients with childbearing potential should use one of the following contraceptives methods: intrauterine devices, barrier methods and tubal ligation

Exclusion Criteria:

* Colorectal cancer without bleeding evidences
* Pregnancy or lactation
* Use of hormonal contraceptives or treatments with sexual hormones in general
* Patients with other illnesses not adequately controlled such as congestive heart failure, arterial blood pressure, unstable angina, severe cardiac arrhythmia, thromboembolic disease, diabetes 1 or 2, any hidden coronary disease determined by previous assessments
* Psychiatric diseases implying patient incompetence
* Known hypersensitivity to desmopressin or vasopressin
* Severe von Willebrand disease (vWD)(defined by vWF<10% Ui/dl) or 2B vWD (defined by increased platelet agregation induced by ristocetin at low concentration) or hemophilia A or B carriers
* History of seizures
* Renal insufficiency (Creatinine clearance < 50 ml/min), hyponatremia (serum sodium lower than the lower limit of normality-UNL)or previous history of hyponatremia
* Syndrome of inappropriate antidiuretic hormone secretion (SIADH)
* Positive serology for hepatitis B, C or known human immunodeficiency virus (HIV) infection
* Known liver disease (cirrhosis, liver enzymes greater than or equal to 1.5 times the upper limit of normality or total bilirubin greater than or equal to 1.5 times the upper limit of normality
* Active infections wich, according to the investigator judgement, coud interfere with patient safety
* Other malignancies, with the exception of basal cell carcinoma, in situ cervical carcinoma, or any other tumour adequately treated and with a disease-free period greater than or equal to 5 years
* Patients receiving or having received other investigational drugs 30 days prior to study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Presence or absence of grade 3 or 4 adverse events related to the study drug, in a maximum of 2 out of 6 patients assessed in each dose level. | Up to one week after the administration of the first dose
  A total of 6 groups with 3 patients each, with different dose ranges and dosing schedules will be assessed.
  The number of patients in each group with grade 3 or 4 adverse events, including clinical or analytical findings, will be determined in order to stablish the maximum tolerated dose.

SECONDARY OUTCOMES:
Number of patients with grade 3 or 4 local adverse events | Up to one week after the administration of the first dose
  Once the maximum tolerated dose is determined, other 12 patients will be assessed to evaluate safety and tolerability of the study drug when administered as monotherapy.
Number of patients with grade 3 or 4 systemic adverse events | Up to one week after the administration of the first dose
  Once the maximum tolerated dose is determined, other 12 patients will be assessed to evaluate safety and tolerability of the study drug when administered as monotherapy.
Number of withdrawn from treatment | Up to one week after the administration of the first dose
Number of patients with partial or complete response in clinical endpoints | Up to one week after the administration of the first dose
  Clinical endpoints such us rectal bleeding, mucorrhea, evacuatory attempts and rectal pain will be assessed before and after treatment with the study drug.
  Response will be classified as complete or partial response.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Roca, MD, Principal Investigator — Hospital de Gastroenterologia ¨B. Udaondo¨
Locations (2):
- Argentina (2):
  - Hospital de Gastroenterologia ¨B.Udaondo¨, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Oncología "Alexander Fleming", Ciudad Autónoma de Buenos Aires, Buenos Aires

REFERENCES:
- [Derived] Iseas S, Roca EL, O'Connor JM, Eleta M, Sanchez-Luceros A, Di Leo D, Tinelli M, Fara ML, Spitzer E, Demarco IA, Ripoll GV, Pifano M, Garona J, Alonso DF. Administration of the vasopressin analog desmopressin for the management of bleeding in rectal cancer patients: results of a phase I/II trial. Invest New Drugs. 2020 Oct;38(5):1580-1587. doi: 10.1007/s10637-020-00914-5. Epub 2020 Mar 12. PMID 32166534